CLINICAL TRIAL: NCT06045910
Title: A Cancer Research UK Phase I/II Trial of ALETA-001 in Participants Who Have Received an Anti-CD19 CAR T-Cell Therapy for the Treatment of B-cell Malignancies
Brief Title: A Phase I/II Trial of ALETA-001 for the Treatment of Participants With B-cell Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Collaborators: Aleta BioTherapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD/23/001; IRAS ID: 1007028 (Other: IRAS)
Record Dates: First submitted 2023-08-15; First posted 2023-09-21 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, B-Cell; Large B-cell Lymphoma
Keywords: Neoplasms; Immunotherapy, Adoptive; Receptors, Chimeric Antigen; Receptors, Antigen, T-Cell; Antigens, CD19
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, B-Cell; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safety Lead-In Phase (Experimental)
  Interventions: Drug: ALETA-001
- Dose Expansion Phase (Experimental)
  Interventions: Drug: ALETA-001

INTERVENTIONS:
Drug: ALETA-001 — ALETA-001 will be administered intravenously (IV) every two weeks.

SUMMARY:
This is a Phase I/II multicentre, open-label trial designed to evaluate the efficacy, safety, tolerability, timing of administration and pharmacokinetics (PK) of a novel chimeric antigen receptor (CAR) T-cell engager, ALETA-001, administered by intravenous (IV) infusion as a single agent every 2 weeks in participants with B-cell malignancies post CD19 CAR T-cell therapy. This first in human study is divided into 2 parts: a safety lead-in phase (Phase I) and a dose expansion phase (Phase II). Different dose levels of ALETA-001 and timing of administration will be evaluated in Phase I in order to define a recommended dosing level and time of administration for Phase II. Phase II will further evaluate the safety, PK and therapeutic activity of ALETA-001.

ELIGIBILITY:
Inclusion Criteria:

For all participants

Criteria to be met prior to enrolment in the trial:

* Aged 16 years or over.
* Written (signed and dated) informed consent and be capable of co-operating with ALETA-001 administration and follow-up.
* Confirmed diagnosis of B-cell NHL according to World Health Organization (WHO) 2016 criteria.
* Eastern Cooperative Oncology Group performance status of 0, 1 or 2.
* Biochemical indices within protocol specified ranges.

Cohort Specific Inclusion criteria (for Phase I Cohorts A & B) Criteria to be met prior to enrolment in the trial.

* Histologically confirmed diagnosis of relapsed/refractory LBCL or MCL.
* Have received an approved anti-CD19 CAR T-cell therapy.
* Objectively evaluable or measurable disease at 4 weeks (±1 week) post CAR T, which demonstrates:

  * inadequate or incomplete response (PR or SD), or
  * PD if there is a reasonable expectation of deriving benefit from trial treatment, or
  * initial response followed by relapse within 9 months assessed according to Lugano Criteria.
* Haematological indices within protocol specified ranges.

Cohort Specific Inclusion criteria (for Phase I Cohorts C & D) Criteria to be met prior to lymphodepleting chemotherapy for CAR T therapy.

* Histologically confirmed diagnosis of relapsed/refractory LBCL or MCL.
* Approved by the UK national CAR T Clinical Panel (NCCP) to receive an approved anti-CD19 CAR T-cell therapy.
* Haematological indices within protocol specified ranges.
* Adequate cardiac function within protocol specified ranges with no clinical symptoms or signs of heart failure.
* Resting O2 saturation of ≥92% on room air.

Eligibility for participants in Phase II of the trial will depend on timing of administration of ALETA-001 which will be recommended by the Safety Review Committee (SRC).

Exclusion Criteria for all participants:

* Active or previous malignancies of other types that, in the opinion of the Investigator, should exclude the participant. Exceptions include adequately treated cone biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin and patients with asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy or who require only hormonal therapy and have had normal prostate specific antigen for >1 year prior to the start of therapy. Cancer survivors, who have undergone potentially curative therapy for a prior malignancy, have no evidence of that disease for 2 years or more and are deemed at negligible risk for recurrence, are eligible for the trial.
* Any ongoing toxic manifestation of previous anti-cancer treatment that, in the opinion of the Investigator, should exclude the participant.
* Ongoing need for systemic immunosuppressive therapy other than replacement dose of corticosteroids. Intermittent topical, inhaled or intranasal corticosteroids are permitted.
* Presence of active infections and/ or inflammatory disease requiring active management.
* Documented current central nervous system involvement by lymphoma.
* Women of childbearing potential (or are already pregnant or lactating) unless willing to adhere to protocol-defined contraceptive requirements.
* Male patients with partners of childbearing potential unless willing to adhere to protocol-defined contraceptive requirements.
* Major thoracic or abdominal surgery from which the participant has not yet recovered.
* At high medical risk because of non-malignant systemic disease including active uncontrolled infection.
* Hypersensitivity to any of the ingredients/excipients in ALETA-001.
* Participation in another interventional clinical trial, whilst taking part in this trial of ALETA-001. Participation in an observational trial or interventional clinical trial that does not involve administration of an IMP and that would not place an unacceptable burden on the participant, in the opinion of the Investigator and CDD, would be acceptable.
* Participants with any congenital or acquired immunodeficiency syndrome or who are receiving immunosuppressive therapy (including any dose of systemic corticosteroids), or who are immunosuppressed post organ transplant. However, participants receiving inhaled corticosteroids and participants with a history of allergy (other than anaphylaxis) are eligible, as are participants with a history of autoimmune disease.
* Any other condition that, in the Investigator's opinion, would mean that the trial is not in the best interests of the participant.
* Concurrent radiotherapy (except for palliative reasons).

Cohort specific exclusion criteria prior to enrolment in the trial (for Phase I

Cohorts A & B):

* Participants who have received any other systemic anti-cancer treatment post-CAR T.
* Potential participants who experienced any of the following because of the initial CAR T treatment:

  * Grade 4 CRS or ICANS post CAR T infusion.
  * Grade ≥3 CRS or ICANS persisting beyond 7 days despite optimal therapy.
  * Any Grade ≥1 CRS or ICANS must have fully resolved.
* Any Grade ≥3 organ toxicity (other than haematologic toxicity) following CAR T infusion must have improved to Grade ≤2 for at least 48 hours prior to ALETA-001 infusion.

Cohort specific exclusion criteria prior to ALETA-001 infusion between Day 10-18 post CAR T-cell infusion (for Phase I Cohorts C & D):

* Grade 4 CRS or ICANS post CAR T infusion.
* Grade ≥3 CRS or ICANS persisting beyond 7 days despite optimal therapy.
* Any Grade ≥2 CRS or ICANS must have improved to Grade ≤1 for at least 48 hours prior to ALETA-001 infusion.
* ECOG performance status ≥3.
* Any Grade ≥3 organ toxicity (other than haematologic toxicity) following CAR T infusion must have improved to Grade ≤2 for at least 48 hours prior to ALETA-001 infusion.
* Any unresolved serious active infection which in the opinion of the Investigator precludes ALETA-001 infusion (ongoing need for IV antimicrobial therapy per se is not an exclusion).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2029-12-21 (Estimated)

PRIMARY OUTCOMES:
Dose level of ALETA-001 and timing of administration for use in Dose Expansion (Safety Lead-in Phase). | Day 1 to Day 28.
  Determine a dose level that is deemed tolerable and timing of administration based on available safety and pharmacodynamic data.
Number of Participants who experience dose limiting toxicities (DLTs). | Up to Day 28.
  DLTs will be assessed up to Day 28 and are defined as toxicities that meet pre-defined severity criteria and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, intercurrent illness, or concomitant medications that occurs within the 28 days of the first dose of ALETA-001.
Number of Participants who experience Grade 3, 4 or 5 related adverse event (AEs). | Safety data will be collected from the time of informed consent until 95 days after the last dose of ALETA-001. The average time from consent to the end of follow up will be presented.
  Related AEs are those considered by the investigator to be possibly, probably or highly probably related to ALETA-001. Events of cytokine release syndrome (CRS) and immune effector cell associated neurotoxicity (ICANS) are graded according to the American Society for Transplantation and Cellular Therapy grading criteria. All other AEs are graded according to the Common Terminology Criteria for AEs (CTCAE) Version 5.0.
Best Overall Response (Dose Expansion Phase). | Radiological assessment from within 28 days before starting ALETA-001 and up to 12 months after.
  Best Overall Response according to Lugano criteria (Cheson, Journal of Clinical Oncology, 2014), the number of participants taking part in the Dose Expansion Phase with best overall response of complete response (CR), partial response (PR), no response or stable disease (SD/NR), and progressive disease (PD).
Progression-Free Survival (PFS) (Dose Expansion Phase). | From date of first dose of ALETA-001 up to 12 months.
  Median PFS measured from first dose of ALETA-001 to date of progression according to Lugano criteria or date of death without a previous progression recorded.
Time to Progression (TTP) (Dose Expansion Phase). | From date of first dose of ALETA-001 up to 12 months.
  Median TTP measured from first dose of ALETA-001 to date of progression according to Lugano criteria. Participants who die without recorded progression will be censored.
Overall Survival (OS) (Dose Expansion Phase). | Follow-up until end of trial, estimated to be up to 48 months.
  Median OS measured from first dose of ALETA-001 to date of death due to any cause or to the date of censoring at the last time the participant was known to be alive.

SECONDARY OUTCOMES:
Best Overall Response (Safety Lead-in Phase). | Radiological assessment from within 28 days before starting ALETA-001 and up to 12 months after.
  Best Overall Response according to Lugano criteria, the number of participants taking part in the Safety Lead-in Phase with best overall response of complete response (CR), partial response (PR), no response or stable disease (SD), and progressive disease (PD).
Progression-Free Survival (PFS) (Safety Lead-in Phase). | From date of first dose of ALETA-001 up to 12 months.
  Median PFS measured from first dose of ALETA-001 to date of progression according to Lugano criteria or date of death without a previous progression recorded.
Time to Progression (TTP) (Safety Lead-in Phase). | From date of first dose of ALETA-001 up to 12 months.
  Median TTP measured from first dose of ALETA-001 to date of progression according to Lugano criteria. Participants who die without recorded progression will be censored.
Overall Survival (OS) (Safety Lead-in Phase). | Follow-up until end of trial, estimated to be up to 48 months.
  Median OS measured from first dose of ALETA-001 to date of death due to any cause or to the date of censoring at the last time the participant was known to be alive.
Maximum observed serum concentration (Cmax) of ALETA-001. | Day 1 to Day 7.
  Measurement of Cmax of ALETA-001 as appropriate.
Terminal elimination half-life (t1/2) of ALETA-001. | Day 1 to Day 7.
  Measurement of t1/2 of ALETA-001 as appropriate.
Area under the concentration-time curve (AUC) of ALETA-001. | Day 1 to Day 7.
  Measurement of AUC of ALETA-001 as appropriate.
Volume of distribution (Vss) of ALETA-001. | Day 1 (before first ALETA-001 infusion) to Day 7.
  Measurement of Vss of ALETA-001 as appropriate.
Clearance (CL) of ALETA-001. | Day 1 to Day 7.
  Measurement of CL of ALETA-001 as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Sridhar Chaganti, Dr, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (7):
- United Kingdom (7):
  - University Hospital Birmingham NHS Foundation Trust, Birmingham
  - Cambridge University Hospitals, Cambridge
  - St James's University Hospital, Leeds
  - University Hospital London Hospital, London
  - Manchester Royal Infirmary, Manchester
  - The Christie Hospital, Manchester
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified patient data that underlie the results reported will be shared with researchers whose proposed use of the data is approved by a review committee of the Sponsor.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All requests made within 5 years from the end of trial will be considered; requests made subsequently will be considered where possible.
Access Criteria: When a request has been approved, Cancer Research UK will provide access to the de-identified individual patient-level data and appropriate supporting information. A signed Data Sharing Agreement must be in place before accessing requested information. Requests should be submitted to drugdev@cancer.org.uk.